CLINICAL TRIAL: NCT05180617
Title: Feasibility of Music Therapy, Neural Processing and Reduction of Craving in Community Substance Misuse Treatment Services (CSMTS)
Brief Title: Feasibility of Music Therapy in Community Substance Misuse Treatment Services
Acronym: CRAVEMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Westminster Drug Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDPARU22
Record Dates: First submitted 2021-12-03; First posted 2022-01-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-01

CONDITIONS: Substance Use Disorders
Keywords: Addiction; Craving; music therapy; mental health; neural dynamics; EEG; Feasibility; emotion processing; drug memory
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Psychological Well-Being | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual music therapy (IMT) (Experimental): After baseline measures, each Participant will receive 6 x 1 weekly hour of music therapy. During music therapy the participants will be interacting both musically and verbally with the therapist.
  Participants will be provided with both acoustic and electronic instruments to be able to improvise with the therapist. In addition, IMT participants will be provided with the opportunity to compose and write songs, take part in preferred music lyric analysis, sing and discuss/talk with the therapist.
  During session 2 and 5 EEG hyperscanning of therapist and patient will be applied.
  All 5 IMT participants will do the same pre-post intervention test battery.
  Interventions: Behavioral: Music Therapy
- Group music therapy (GMT) (Experimental): During 6 x 1 weekly hour of GMT, 5 participants will be invited to take part in a range of group music making activities.
  Participants will be provided with both acoustic and electronic instruments to be able to improvise within the group setting. In addition, GMT participants will be provided with the opportunity to compose and write songs as a group, take part in preferred music lyric analysis, sing and take part in group discussions.
  All 5 GMT participants will do the same pre-post intervention test battery.
  Interventions: Behavioral: Music Therapy
- Control Group (No Intervention): CG will receive standard treatment, which includes key work sessions, other group work programmes and clinical support (e.g. prescribing).
  All 5 CG participants will do the same pre-post intervention test battery.

INTERVENTIONS:
Behavioral: Music Therapy — Music therapy participants will interact both musically and verbally with the therapist and will be given a range of both electronic and acoustic instruments to choose from. Music therapy sessions will be based upon music improvisation, and as such participants are not required to have any previous instrument or other music experience and be invited to improvise freely using the instruments. The music therapist will accompany participants in the improvisation. This provides participants with an opportunity to connect with emotions and feelings connected to hidden psychic material. Following improvisations, the therapist and client will identify these moments of interest which can be further explored either verbally or through further improvisation. The music created within sessions will be recorded and participants can take a copy of the recordings home and it will be used in the therapeutic monitoring and analysis of sessions.
  Arms: Group music therapy (GMT); Individual music therapy (IMT)

SUMMARY:
Music Therapy (MT) has been shown to improve several symptoms experienced by people with Substance Use Disorder (SUD), such as depressive and anxiety symptoms, as well as negative emotions. Particularly, a recent Cochrane review reported craving reduction as a main outcome for MT delivered to SUD participants. The possible mechanism(s) of therapeutic change is yet to be identified and future randomized control trials applying neuroscience research methods may help doing so. However, there is a significant lack of studies investigating those effects in a specific cohort of out-patients on prescription medicine from Community Substance Misuse Treatment Services (CSMTS). This research project aims to evaluate the acceptability and feasibility of MT and the applied test battery in CSMTS for a future Randomised Controlled Trails (RCT).

Fifteen participants from a CSMTS will take part in a three-arm randomized non-blind controlled trial. 5 participants will receive 6 weekly individual music therapy sessions (IMT), 5 participants will receive 6 weekly group music therapy (GMT) sessions and 5 participants will act as a control group (CG) receiving treatment as usual (TAU). IMT and GMT participants will continue to receive TAU by the CSMTS. The CG will have the opportunity to receive MT as well, after the end of the study.

Regarding the feasibility of the service implementation, the investigators will evaluate participant satisfaction and implement a focus group following the final session to collect feedback and evaluation on acceptability of the intervention from both participants and staff. Moreover, retention in treatment and completion rates will be measured after the end of the MT sessions.

Furthermore, based on previous research and the theoretical basis of MT interventions, the investigators aim to explore the effects of MT on craving, substance use, symptoms of depression and anxiety, and inhibitory control in people with SUD. Changes in the brain correlates of the abovementioned symptoms will be investigated as well as how music and emotion are processed in the brain during MT. The investigators will collect subjective and objective baseline measurements and compare them against post-treatment measurements. Some variables of interest will be measured by Electroencephalography (EEG) which is a non-invasive technique to record electrical brain activity.

The study will take place in a Westminster Drug Project provided community-based integrated adult substance misuse service in London. Participants will be recruited from service users receiving treatment at this service.

DETAILED DESCRIPTION:
This feasibility research project seeks to support individuals receiving treatment from a Community Substance Misuse Treatment Service (CSMTS) in reducing symptoms of craving, anxiety, depression and negative emotion through either group or individual music therapy sessions.

To test the feasibility of the implementation into CSMTS and the application of a test battery including self-report, interviews and physiological measures, a total of 15 adult participants will be randomly allocated to three arms of the study. The participants will receive either Group Music Therapy (GMT) alongside Standard Treatment (ST), Individual Music Therapy (IMT) alongside Standard Treatment or Standard Treatment only. Music therapy (MT) sessions will provide an opportunity for participants to interact musically with the music therapist using acoustic and electronic instruments. During the study, participants will be asked to complete questionnaires and behavioural measures and participate in electroencephalography recordings.

For SUD participants, the duration of their direct involvement with the research will be 9 weeks. Additional data will be gathered by the research team at 1 month post-intervention: this will not require participant involvement as this data will be captured from the Westminster Drug Project's (WDP) patient database.

Prior to and following the research intervention, participants have been (and will be) consulted and given the opportunity to provide feedback on the research design. Where appropriate, changes were made to the research procedures to reflect this feedback.

Propositions.

Previous studies found therapeutic effects of MT on several substance misuse - related outcomes such as depressive symptoms, anxiety, negative emotions (i.e. anger) and subjective feeling of craving. However, there's a lack of studies investigating and adding explanatory value to these outcomes in CSMTS.

Based on previous research and the theoretical basis of MT interventions, the investigators aim to explore the effects of MT in addition to ST versus ST alone.

The investigators propose that this MT intervention will a) be feasible and acceptable for individuals receiving community-based substance misuse treatment, b) lead to a decrease in symptoms of anxiety, depression and craving; c) improve treatment outcomes for those in community substance misuse treatment services; d) improve inhibitory control, potentially correlating with changes in craving state.

Furthermore, the investigators will explore the feasibility of measuring neural correlates of moments of therapeutic interest regarding craving, strong emotion and therapeutic relationship during IMT sessions with EEG Hyperscanning and audio-visual monitoring in sessions 2 and 5. The investigators expect moments of strong emotion and increased therapeutic relationship to occur more often in the later session. The investigators will record and analyse participants' engagement with electronic music production instruments (EMPI) and acoustic instruments. Hyperscanning, and high-quality session recordings will allow analysing continuous data of contextualised events and moments of therapeutic interest during IMT.

Research methodology.

To approach these propositions the research team has identified that a feasibility/pilot study employing three study arms would be most appropriate. The study will involve the recruitment of 15 adult participants receiving treatment for substance misuse and are experiencing self-reported symptoms of depression/anxiety.

The study is designed as a three-armed study with group 1 receiving 6 weekly sessions of Group Music Therapy (GMT) and ST, group 2 receiving 6 weekly sessions of Individual Music Therapy (IMT) and ST and group 3, which is a control group (CG), receiving 6 weeks of ST only.

In addition to a post intervention focus group session with MT participants, the investigators will recruit a Staff Group (SG) of 4-8 WDP staff who will participate in a focus group after both sets of MT have been delivered. The staff focus group will explore the feasibility of MT from a number of perspectives, including those involved in the set-up of the MT sessions.

Research duration.

The duration of this research is outlined to be a period of 6 months. Participants will be committing to attend 6 weekly music therapy sessions, a focus group (consisting of participants from IMT and GMT) to gather participant's feedback on feasibility and accessibility, and only for GMT participants, an individual debriefing interview with the therapist.

In addition to this, those considering participating will have an opportunity, prior to volunteering, to meet with the research team and take part in a workshop where the research team will describe and demonstrate the process of MT, providing an opportunity for potential participants to ask questions and provide feedback. This introductory session will be in addition to the 8-week commitment the investigators are seeking from participants.

While participants will be committing for 8 weeks, the research team will carry out further investigations at week 11 (1 month post intervention).

Recruitment.

Recruitment will be carried out by advertising the project in the service and by WDP staff identifying eligible service users through WDP's case management system. Service users will be asked by their keyworker to provide the information sheets and informed consent form. For those that have not been identified through the case management system but approached by their keyworker, the keyworker or service admin will ascertain eligibility through the case management system and in the keyworker session. If eligible, the information sheets and informed consent form will be handed out.

The research team has already consulted with 7 service users, presented the design and received positive feedback on the current design. The research team will seek further input from service users through WDP's service user consultation process and hold a presentation of the research project within the service to interested service users. This presentation will seek to aid recruitment and provide further information about the project and what participation will involve as well as give interested service users a chance to ask the research team questions.

Those service users who are interested in being considered for the study will be asked to complete the consent form and hand this to either their key-worker or a member of WDP's Innovation and Research research team.

Upon their recruitment, each of the 15 participants will be assigned a unique, randomly generated number to anonymise their personal information.

The investigators will also recruit up to 8 WDP staff members, who were involved in the implementation of the intervention, to a single focus group after the music therapy intervention is complete. The Staff group (SG) will not receive music therapy.

Research Procedure.

Following recruitment, participants will be randomly allocated to one of the three research groups: group 1 receiving GMT and ST, group 2 receiving IMT and ST and group 3 receiving ST only.

The planned schedule will be:

Week 1: GMT, IMT and CG baseline (pre-intervention) measures at time point 1 (TP1).

Weeks 2-7: GMT and IMT receive 6 weekly MT sessions plus ST; GMT and IMT pre-post session measures; CG receives ST only; IMT only: EEG Hyperscanning during Session 2 (week 3) and session 5 (week 6) and post session interview and questionnaire

Week 8: GMT, IMT and CG post-intervention measures and participant satisfaction survey at time point 2 (TP2)

Week 9: Feasibility Focus groups for SG, GMT and IMT; Individual debriefing interview with therapist for GMT participants only

Week 11: (1 months post intervention): all groups (excluding staff group) will have retention in treatment, treatment engagement and completion rate taken from WDP's Case management system

ELIGIBILITY:
Inclusion Criteria:

* Service users in structured treatment for drug and/or alcohol misuse,
* Aged 18-65
* Reporting / Self-reporting symptoms of depression and/or anxiety.
* Service users will need to be deemed suitable to take part in a group / individual setting by their key workers.
* Right-handedness

Exclusion Criteria:

* Service users on medication for depression or anxiety,
* Services users who are currently receiving treatment as part of a Drug Rehabilitation Requirement (DRR) or Alcohol Treatment Requirement (ATR).
* Service users who are unable to provide informed consent due to a lack of mental capacity,
* Service users with little/no understanding of spoken English.
* Service users with a brain injury or history of epilepsy.
* Left-Handedness
* Mixed-Handedness
* Not registered with a General Practitioner (GP) / unable to provide GP details

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Retention in Treatment 1 (Attendance Sheet) | up to 6 weeks
  Retention in treatment will be assessed through an attendance sheet to be completed by the music therapist and the participants receiving Group Music Therapy (GMT) and Individual Music Therapy (IMT) after each session (6 sessions). In this way, participants' feedback will be taken throughout the treatment process.
Acceptability of Treatment 1 (Participant Satisfaction Survey) | Post-Intervention Measure: at week 8
  Regarding the feasibility of the service implementation, the investigators will evaluate participant satisfaction and implement a focus group following the final session to collect both participants and staff feedback and evaluation.
  A Participant Satisfaction Survey will be conducted at week 8 (end of treatment) to the 10 participants receiving group music therapy (GMT) and individual music therapy (IMT).
Acceptability of treatment 2 (Focus Groups) | Post-Intervention Measure: at week 9
  Regarding the feasibility of the service implementation, the investigators will evaluate participant satisfaction and implement a focus group following the final session to collect both participants and staff feedback and evaluation.
  FOCUS GROUPS (FG). The feasibility of the music therapy intervention will be assessed with FG after the intervention.
  FG 1 will consist of individual and group music therapy members ; FG 2 will consist of 4 WDP service staff members attending a single focus group to explore staff perspectives on MT.
Retention in Treatment 2 (Treatment Status) | 1-month post-intervention: at week 11
  The treatment status from participants receiving Individual Music Therapy (IMT), Group Music Therapy (GMT) and Standard Treatment (ST) will be collected by WDP's case management system and will provide information about retention in treatment, treatment engagement and completion rate taken from WDP's Case management system

SECONDARY OUTCOMES:
The Brief Substance Craving Scale (BSCS) | At baseline (week 1) and end of treatment (week 8)
  The Brief Substance Craving Scale (BSCS) is a multi-item subjective measure to assess changes in craving symptoms experienced over a 24-h period. It ranges from 0-12, with 12 indicating the highest level of craving.
Craving Thermometer VAS | up to 6 weeks
  The craving thermometer is a visual analogue scale (VAS) type of measure that allows a quick one-click estimate of the instantaneous subjective feeling of craving (from 0-100). Participants will be asked to indicate their level of craving by responding to the question: "Please, rate how strong your drug craving is right now by putting a mark on the line going from not craving at all to the most ever". Participants will simply read the question and evaluate their subjective feeling of instantaneous craving by putting a mark at any level on the horizontal line. Then, responses will be recorded as a 0 to 10 score (including decimal numbers). The Craving Thermometer will be administered before and after each MT session.
The Treatment Outcome Profile (TOP) | At baseline (week 1) and end of treatment (week 8)
  The Treatment Outcome Profile (TOP) is a multi-item subjective measure to assess changes in substance use, days of primary substance used, usage of primary substance per day, physical wellbeing, mental wellbeing and overall quality of life compared to a baseline measurement.
The Patient Health Questionnaire (PHQ-9) | At baseline (week 1) and end of treatment (week 8)
  The Patient Health Questionnaire (PHQ-9) is a multi-item questionnaire to assess changes in depressive symptoms.
The Generalised Anxiety Disorder Assessment (GAD-7) | At baseline (week 1) and end of treatment (week 8)
  The Generalised Anxiety Disorder Assessment (GAD-7) is a multi-item subjective measure to assess changes in anxiety symptoms.
Resting-state EEG frontal alpha asymmetry (FAA) | At baseline (week 1) and end of treatment (week 8)
  Resting-state EEG frontal alpha asymmetry (FAA) will be a measure to evaluate the neural correlates of depressive symptoms.
Resting-state EEG frontal midline theta (FMT) | At baseline (week 1) and end of treatment (week 8)
  Resting-state EEG frontal midline theta (FMT) will be a measure to evaluate the neural correlates of anxiety symptoms.
Resting-state EEG beta frequency band | At baseline (week 1) and end of treatment (week 8)
  Resting-state EEG variation of the beta frequency band will be a measure to evaluate the neural correlates of craving.
Go/No-Go Event-Related Potentials (ERPs) task | At baseline (week 1) and end of treatment (week 8)
  A behavioural measure (accuracy) during a Go/No-Go task and EEG ERP P3 amplitude will be collected to assess inhibitory control in participants allocated to IMT, GMT and ST.
EEG Hyperscanning | At week 3 and week 6
  In the IMT arm of the study Dual-EEG (EEG hyperscanning) will be measured from the therapist and from the participant to test the feasibility of using the hyperscanning to study the mechanism of change and potentially to collect data on the time course of emotional processing and therapeutic relationship. The EEG hyperscanning data will be collected throughout the music therapy sessions 2 and 5.
Dual EEG resting-state Frontal Alpha Asymmetry | At week 3 and week 6
  In the IMT arm of the study 5-minutes of Dual EEG resting-state data from therapist and patient before the beginning and at the end of therapy session 2 and 5 will be recorded.
  This will allow to assess pre-post session changes in the neural correlates of depressive symptoms with Frontal Alpha Asymmetry.
Dual EEG resting-state Frontal Midline Theta | At week 3 and week 6
  In the IMT arm of the study 5-minutes of Dual EEG resting-state data from therapist and patient before the beginning and at the end of therapy session 2 and 5 will be recorded.
  This will allow to assess pre-post session changes in the neural correlates of anxiety symptoms with Frontal Midline Theta.
Dual EEG resting-state Beta waves | At week 3 and week 6
  In the IMT arm of the study 5-minutes of Dual EEG resting-state data from therapist and patient before the beginning and at the end of therapy session 2 and 5 will be recorded.
  This will allow to assess pre-post session changes in the neural correlates of craving symptoms with beta waves.
Semi-structured interview | At week 3 and week 6
  After session 2 and session 5 in the IMT arm of the study a semi-structured interview will be conducted to explore moments of therapeutic interest. These moments will be selected by importance and emotional relevance. Participants may also report verbally any craving related experience. Moments of interest will be identified and located in the recording session. These reports and their timestamp of occurrence will be entered into a therapy event log. The interview will potentially help to select and identify therapeutically important moments: defined as moments of interest (MOI). This is important to describe a narrative of the therapeutic change process and to analyse EEG event-related temporal dynamics during MOI as compared to moments of non-interest (MONI).
  This semi-structured interview will also be conducted to explore participants' perspective and experience of using music technology in a music therapy intervention.
Helping Alliance Questionnaire - II (HAQ-II) | At week 3 and week 6
  The Helping Alliance Questionnaire - II (HAQ-II) will be completed by both the therapist and the client. The HAQ-II is a 19 item questionnaire measuring the quality of the therapist-patients relationship on a scale ranging from 1-6, with 6 indicating the highest helping alliance rating.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Murtagh, Principal Investigator — WDP; Jorg C Fachner, PhD, Study Director — Anglia Ruskin University
Locations (1):
- Westminster Drug project, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fachner, J. (2017). Retraining of Drug Reward, Music Cues and State-dependent Recall in Music Therapy. Music and Medicine, 9(1), 8-14.
- [Background] Ridder HM and Fachner J. (2016) Objectivist case study research. Single-subject and small-n research. In: Wheeler B and Murphy K (eds) Music Therapy Research. 3 ed. Dallas: Barcelona Publishers, 291-302.
- [Result] Albornoz, Y. (2011). The effects of group improvisational music therapy on depression in adolescents and adults with substance abuse: a randomized controlled trial. Nordic Journal of Music Therapy, 20, 208-224.
- [Result] Cevasco AM, Kennedy R, Generally NR. Comparison of movement-to-music, rhythm activities, and competitive games on depression, stress, anxiety, and anger of females in substance abuse rehabilitation. J Music Ther. 2005 Spring;42(1):64-80. doi: 10.1093/jmt/42.1.64. PMID 15839734
- [Result] Eshaghi Farahmand, S. R., Ahadi, H., Kalhornia Golkar, M., & Sedaghat, M. (2020). Comparison of the Effectiveness of Music Therapy and Cognitive Behavioral Therapy on Quality of Life, Craving and Emotion Regulation in Patients Under Methadone Maintenance Therapy. Iranian Journal of Psychiatry and Clinical Psychology, 26(2), 170-187.
- [Result] Silverman, M. J. (2019). Effects of group-based educational songwriting on craving in patients on a detoxification unit: A cluster-randomized effectiveness study. Psychology of Music, 47(2), 241-254.
- [Result] Hohmann L, Bradt J, Stegemann T, Koelsch S. Effects of music therapy and music-based interventions in the treatment of substance use disorders: A systematic review. PLoS One. 2017 Nov 15;12(11):e0187363. doi: 10.1371/journal.pone.0187363. eCollection 2017. PMID 29141012
- [Result] Fachner JC, Maidhof C, Grocke D, Nygaard Pedersen I, Trondalen G, Tucek G, Bonde LO. "Telling me not to worry..." Hyperscanning and Neural Dynamics of Emotion Processing During Guided Imagery and Music. Front Psychol. 2019 Jul 25;10:1561. doi: 10.3389/fpsyg.2019.01561. eCollection 2019. PMID 31402880
- [Result] Kamarajan C, Porjesz B, Jones KA, Choi K, Chorlian DB, Padmanabhapillai A, Rangaswamy M, Stimus AT, Begleiter H. Alcoholism is a disinhibitory disorder: neurophysiological evidence from a Go/No-Go task. Biol Psychol. 2005 Jul;69(3):353-73. doi: 10.1016/j.biopsycho.2004.08.004. Epub 2004 Nov 21. PMID 15925035
- [Result] Huang Y, Mohan A, De Ridder D, Sunaert S, Vanneste S. The neural correlates of the unified percept of alcohol-related craving: a fMRI and EEG study. Sci Rep. 2018 Jan 17;8(1):923. doi: 10.1038/s41598-017-18471-y. PMID 29343732
- [Result] Ghetti C, Chen XJ, Brenner AK, Hakvoort LG, Lien L, Fachner J, Gold C. Music therapy for people with substance use disorders. Cochrane Database Syst Rev. 2022 May 9;5(5):CD012576. doi: 10.1002/14651858.CD012576.pub3. PMID 35532044
- [Result] Carter, T.E., Panisch, L.S. A Systematic Review of Music Therapy for Psychosocial Outcomes of Substance Use Clients. *Int J Ment Health Addiction* **19,** 1551-1568 (2021). https://doi.org/10.1007/s11469-020-00246-8
- [Derived] Fachner J, Maidhof C, Murtagh D, De Silva D, Pasqualitto F, Fernie P, Panin F, Michell A, Muller-Rodriguez L, Odell-Miller H. Music therapy, neural processing, and craving reduction: an RCT protocol for a mixed methods feasibility study in a Community Substance Misuse Treatment Service. Addict Sci Clin Pract. 2023 May 27;18(1):36. doi: 10.1186/s13722-023-00385-y. PMID 37245018